CLINICAL TRIAL: NCT05167695
Title: Maintaining Behavior Change: An Evaluation of a Habit-based Sleep Health Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Allison Harvey, Professor of Clinical Psychology, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-06-14409
Record Dates: First submitted 2021-11-29; First posted 2021-12-22 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Circadian Dysregulation
Keywords: Habits; Circadian; Sleep; transdiagnostic; Intervention
MeSH Terms: conditions — Chronobiology Disorders; Habits

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Habit-based Sleep Health Intervention (HABITs) (Experimental): Participants in this condition participate in the HABITs intervention which includes 3x50-minute weekly sessions followed by 6x30-minute weekly sessions.
  Participants in this group will not receive the texts discussed below.
  Interventions: Behavioral: Habit-based Sleep Health Intervention
- Habit-based Sleep Health Intervention plus text messages (HABITs+texts) (Experimental): Participants in this condition participate in the HABITs intervention which includes 3x50-minute weekly sessions followed by 6x30-minute weekly sessions.
  Additionally, participants in this group will receive the text messaging intervention.
  Interventions: Behavioral: Habit-based Sleep Health Intervention; Behavioral: Text messaging intervention

INTERVENTIONS:
Behavioral: Habit-based Sleep Health Intervention — A novel low-cost approach derived by leveraging the science of habit formation
Behavioral: Text messaging intervention — In addition to the Habit-based Sleep Health Intervention, the participants will also receive the text messaging intervention.
  Arms: Habit-based Sleep Health Intervention plus text messages (HABITs+texts)

SUMMARY:
The study will test a sleep-health intervention that leverages the science on habit formation. It will evaluate if adding a text messaging intervention improves habit formation. The participants will be 18-30 years old.

DETAILED DESCRIPTION:
The study will test a sleep-health intervention that leverages the science on habit formation. Additionally, the investigators will evaluate whether adding a text messaging intervention improves habit formation. The participants will be 18-30 years old. This is a distinct developmental period in which priorities shift toward self-sufficiency and personal responsibility, which are supported by developing adaptive habits.

Main Aim. To evaluate if adding a text messaging intervention, derived from learning theory, to HABITs improves the utilization of sleep health behavior and improves sleep and circadian outcomes and functioning in the five health-relevant domain outcomes in the short (post-treatment) and longer term (6 and 12-months later), relative to HABITs without text messaging.

Main Hypothesis. Relative to HABITs, youth in HABITs+Texts will (a) establish stronger sleep health behavior habits, (b) report utilizing more sleep health behaviors and (c) exhibit improved sleep and circadian functioning and lower health-relevant risk. These effects will be observed at post-treatment as well as 6 and 12-months later.

Exploratory Aim: To evaluate if the Habit-based Sleep Health Intervention ('HABITs') is associated with an improvement in the utilization of sleep health behavior, an improvement in sleep and circadian outcomes and an improvement in functioning in the five health-relevant domain outcomes in the short (post-treatment) and longer term (6 and 12-months later), relative to baseline.

Exploratory Hypothesis. Combining across the HABITs and HABITs+Texts treatment arms, receiving either intervention will be associated with (a) improved sleep health behavior habits, (b) more utilization of sleep health behaviors, (c) improved sleep and circadian functioning and (d) lower health-relevant risk at post-treatment, 6- and 12-month follow-up, relative to baseline.

Additional exploratory analyses: To examine (a) if sleep health behavior that has become habitual mediates the effects of treatment on improvement in sleep, circadian and health outcomes and (b) if intervention effects are moderated by selected variables (e.g., age, sex, minority group, socioeconomic status (SES), season).

ELIGIBILITY:
Inclusion Criteria:

1. Scoring less than or equal to 26 on the Composite Scale of Morningness OR Mid-point of sleep later than 4:30 AM for 18-24 yo and 3:50 AM for 25-30 yo on work-free/weekend days over the past month OR Night-to-night variation in sleep and wake times across one month of 2 hours or more.
2. 'At risk' in one of the five health domains: the emotional domain, the cognitive domain, the behavioral domain, the physical domain and the social domain. "Risk" is defined as scoring 4 or higher on one item from an adapted version of the Work and Social Adjustment Scale.
3. Age between 18 and 30.
4. English language fluency.
5. Able and willing to give informed assent.
6. If taking medication for sleep, the dose and frequency of use must have been stable for at least 4 weeks.

Exclusion Criteria:

1. Presence of substance abuse/dependence, mental illness, physical illness, suicidality or developmental disorder only if it makes participation in the study unfeasible or if there is a significant risk of harm and/or decompensation if treatment of that comorbid condition is delayed due to participating in this study.
2. Evidence of sleep apnea, restless legs or periodic limb movements during sleep. Youth presenting with provisional diagnoses of any of these disorders will be referred for a non-study polysomnography evaluation and will be enrolled only if the diagnosis is disconfirmed or if the disorder is treated.
3. Night shifter worker where the shift is scheduled between the hours of midnight to 6am > 2 nights per week.
4. Pregnancy or breast-feeding.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Self-Report Automaticity Habits Index integrated with the Utilization Scale | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  16-item; 0-4 scale. Scores can range from 0 to 64 (Higher score means more automaticity in utilization).
Utilization Scale | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  16-item; 0-4 scale. Scores can range from 0 to 64 (Higher score means more utilization).
Composite Sleep Health Score | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  Composite Sleep Health Score which is defined as the sum of scores on 6 sleep health dimensions: Regularity (Midpoint fluctuation), Satisfaction (Sleep quality question on PROMIS-SD), Alertness (Daytime sleepiness question on PROMIS-SRI), Timing (Mean midpoint), Efficiency (Sleep efficiency) and Duration (Total Sleep Time). The Sleep Health Composite was constructed such that higher score indicates better sleep health.
Composite Scale of Morningness | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  Sum of 13-item; Mix of 4-point and 5-point response scale. Scores can range from 13 (extreme evening) to 55 (extreme morning).
Patient-Reported Outcomes Measurement Information System - Sleep Related Impairment (PROMIS-SRI) | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  Sum of 8-items rated on a 5-point response scale. Scores can range from 8 to 40 (Higher score means more Sleep Related impairment)
Patient-Reported Outcomes Measurement Information System - Sleep Disturbance (PROMIS-SD) | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  Sum of 8-items rated on a 5-point response scale. Scores can range from 8 to 40 (Higher score means more Sleep Disturbance)
Adapted version of the Work and Social Adjustment Scale | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  A measure of emotional, cognitive, physical, social and behavioral risk. The 5 items are each rated on a 0-8 scale. The 5 individual item scores will be summed into a total score (range: 0 to 40; Higher score means worse outcome).

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  19-item. First four items are integer responses. The rest of the items are on a 0-3 scale. Creates 7 composite scores, with the sum of the composite scores ranging from 0 to 21. (Higher score means increased severity of difficulty in all sleep area components).
Sleep Diary | Baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  (Not a scale); Night-to-night variability in the mid-point of sleep
Actigraphy | Baseline to 1-week post treatment
  (Not a scale); Night-to-night variability in the mid-point of sleep
Depression, Anxiety, and Stress Scale (DASS) | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  Three subscales-depression, anxiety, stress-of 7 items each, ranging from 0-3 per item. Subscale scores range from 0-21. Final scores are multiplied by two. Higher scores mean worse outcomes. Total score will also be calculated.
Brief Sensation Seeking Scale | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  8-item; 5-point response scale; Scores can range from 8 to 40 (Higher score means higher sensation seeking).
Physical Health Questionnaire | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  Sum of 15-item, 0-2 response scale. Scores can range from 0 to 30 (Higher score means worse physical symptoms)
PROMIS-Cognitive Function | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  6-item; 1-5 response scale. Scores can range from 6-30 (Higher score means better cognitive functioning)
PROMIS-Ability to participate | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  4-item; 1-5 response scale. Scores can range from 4-20 (Higher score means better social functioning)
Ecological Momentary Assessment Composite Risk Score of Functioning - Emotion | Change from baseline to 1-week post treatment
  (Not a scale) Measured via Ecological Momentary Assessment. a 16-item version of the Positive and Negative Affect Schedule will be administered. The Positivity Ratio will also be calculated.
Ecological Momentary Assessment Composite Risk Score of Functioning - Cognitive Domain | Change from baseline to 1-week post treatment
  (Not a scale) Measured via Ecological Momentary Assessment. Concentration, distractedness and focus are rated on a 5 point scale.
Ecological Momentary Assessment (EMA) Composite Risk Score of Functioning - Behavioral Domain | Change from baseline to 1-week post treatment
  (Not a scale) Measured via Ecological Momentary Assessment. The investigators assess eating, caffeine, alcohol, nicotine, marijuana, opioids and prescription and over the counter (OTC) stimulants and sleep aids. Participants will also be asked to list the use of additional psychoactive drugs (e.g. cocaine). The investigators tabulate the average weekly frequency and intake of each substance.
Ecological Momentary Assessment Composite Risk Score of Functioning - Social Domain | Change from baseline to 1-week post treatment
  (Not a scale) Measured via Ecological Momentary Assessment. will assess if the participant is with anyone at the time of the call. Positivity Ratio (see EMA for Emotional Health) will be calculated when the participant is alone, with a family member or with a friend.
Ecological Momentary Assessment Composite Risk Score of Functioning - Physical Domain | Change from baseline to 1-week post treatment
  (Not a scale) Measured via Ecological Momentary Assessment. Physical activity and sedentary behaviors will be assessed.
Self Report Habit Index: Primary habit bundle to build | At the end of the 2nd through last treatment session, which starts 2 to 3 weeks after the beginning of treatment. Also at 1-week post treatment, 6-month follow-up and 12-month follow-up
  6 items rated on 1-5 scale. Scores can range from 1 to 30
Self Report Habit Index: Primary habit bundle to dismantle | At the end of the 2nd through last treatment session, which starts 2 to 3 weeks after the beginning of treatment. Also at 1-week post treatment, 6-month follow-up and 12-month follow-up
  6 items rated on 1-5 scale. Scores can range from 0 to 30

OTHER OUTCOMES:
Adapted version of the Work and Social Adjustment Scale (individual items) | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  A measure of emotional, cognitive, physical, social and behavioral risk. The 5 items are each rated on a 0-8 scale. The 5 individual item scores will be reported separately (range: 0 to 8; Higher score means worse outcome).
Self Report Habit Index: Secondary habit bundle to build | At the end of the 2nd through last treatment session, which starts 2 to 3 weeks after the beginning of treatment. Also at 1-week post treatment, 6-month follow-up and 12-month follow-up
  1 item rated on 1-5 scale. Scores can range from 1 to 5
Self Report Habit Index: Secondary habit bundle to dismantle | At the end of the 2nd through last treatment session, which starts 2 to 3 weeks after the beginning of treatment. Also at 1-week post treatment, 6-month follow-up and 12-month follow-up
  1 items rated on 1-5 scale. Scores can range from 1 to 5
Height | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  (cm)
Weight | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  Pounds (lbs)
Hip circumference | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  (cm)
Waist circumference | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  (cm)
Sleep Diary | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  (Not a scale); Consensus sleep diary variables, including total sleep time, bedtime, and wake-time, calculated separately for weekdays and weekends.
Actigraphy | Change from baseline to 1-week post treatment
  (Not a scale); Sleep parameters, including sleep onset time, sleep offset time, and total sleep time, calculated separately for weekdays and weekends.
Sussex-Oxford Compassion Scale (SOCS) | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  Sum of 20-item, 5-point response scale. Scores can range from 20 to 100 (Higher score means higher compassion for self).
  Sub-scale items included.
Suicidal Behavior Questionnaire - Revised | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  4-item. Total scores can range from 3-18 (Higher Score means higher Suicidal ideation)
  Sub-scale items included.
Alexian Brothers Urge to Self Injure Scale | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  5-item. 0-6 point scale. Total scores can range from 0-30 (Higher Score means higher Suicidal ideation)
State authenticity | Change from baseline to 1-week post treatment, 6-month follow-up and 12-month follow-up
  A measure of state authenticity. The 4 items are each rated on a 1-7 scale. The sum is averaged (range 1-7; higher scores mean more authenticity)
Past month estimates of sleep mid-point workfree days and night-to-night sleep variability | Once at baseline
  Questions to assess mid-point and night-to-night variability eligibility criteria
Sleep Medication Log | Once at baseline
  Questions to assess use of medications
Credibility Expectancy Questionnaire | After the 2nd treatment session, which is 2 to 3 weeks after the beginning of treatment. Again at the post-treatment assessment which is 1-week post treatment
  first 3 items are on a 1-9 scale. The final item is on a 0-100 scale. (Higher score means the treatment was evaluated as more credible).
Adverse Events Checklist | At the 1-week post treatment assessment only
  16 items to assess adverse events experienced during treatment
Proportion of text messages read | At the 1-week post treatment assessment only
  1 item rated from 0% to 100%
Script Elicitation Worksheet | After starting treatment, at the end of the 1st through 3rd treatment session (week 1 through week 3 of treatment)
  (Not a scale); Individualized for each patient, the worksheet includes primary and secondary habit bundles to build and dismantle (e.g., sleep-onset habits, WASO habits, rise-up habits, daytime habits, sleep efficiency habits), and strategy to dismantle primary and secondary habit bundles (e.g., substitution, removing or curtailing, reorganizing)
Proportion of text message prompts participants responded to | After the third treatment session to the ninth and final treatment session (week 3 to week 8)
  (Not a scale) Calculated as the number of times a participant responded to a text prompt, divided by the total number of text prompts sent, and multiplied by 100 to produce a percentage from 0% to 100%. In this trial, the total number of prompts sent to individual participants varied (range: 37 to 105), and the total number of responses from participants ranged from 0 to 76.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Harvey, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California, Berkeley, California, United States

REFERENCES:
- [Derived] Diaz M, Ovalle Patino E, Oliver S, Tiab SS, Salazar N, Song J, Dong L, Sarfan LD, Susman ES, Agnew ER, Gardner B, Harvey AG. Integrating habit science and learning theory to promote maintenance of behavior change: does adding text messages to a habit-based sleep health intervention (HABITs) improve outcomes for eveningness chronotype young adults? Study protocol for a randomized controlled trial. Trials. 2024 Nov 20;25(1):782. doi: 10.1186/s13063-024-08599-4. PMID 39563407